CLINICAL TRIAL: NCT05325489
Title: Comparison Between the Effect of Nebulized Budesonide and Intranasal Budesonide Spray on Children With Adenotonsillar Hypertrophy: A Randomized Controlled Clinical Trial
Brief Title: Comparison of Nebulized Budesonide and Intranasal Budesonide Spray in Children With Adenotonsillar Hypertrophy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Li Shisheng, Associate professor, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LYG2021091
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Snoring; Mouth Breathing
Keywords: adenotonsillar hypertrophy; Nebulization; Intranasal Budesonide Spray
MeSH Terms: conditions — Snoring; Mouth Breathing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebulized Budesonide (Experimental): Drug: budesonide 0.5mg/2ml Pulmicort Respules budesonide inhalation suspension(BIS) once a day (QD) oral montelukast sodium chewable tablets 4mg QD
  Interventions: Drug: Nebulized Budesonide
- Intranasal Budesonide Spray (Active Comparator): Drug: budesonide nasal spray 100μg QD oral montelukast sodium chewable tablets 4mg QD
  Interventions: Drug: Intranasal Budesonide Spray

INTERVENTIONS:
Drug: Nebulized Budesonide — use 0.5mg/2ml Pulmicort Respules BIS QD and oral montelukast sodium chewable tablets 4mg QD
  Arms: Nebulized Budesonide
Drug: Intranasal Budesonide Spray — nasal spray 100μg QD and oral montelukast sodium chewable tablets 4mg QD
  Arms: Intranasal Budesonide Spray

SUMMARY:
Budesonide is one of the most common drugs uesd in children with adenotonsillar hypertrophy. This study aim to evaluate the efficacy of a short course of budesonide inhalation suspension via transnasal nebulization in children with adenotonsillar hypertrophy. The second aim is to compare budesonide inhalation suspension with budesonide aqueous nasal spray in adenotonsillar hypertrophy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children are ≥3 years and ≤10 years, have habitual mouth breathing or snoring, and without current or previous use of any corticosteroids or leukotriene receptor inhibitors within 4 weeks preceding the initial study.

Exclusion Criteria:

* Children with craniofacial, neuromuscular, syndromic, or defined genetic abnormalities; acute upper respiratory tract infection; whose symptoms are not caused by adenotonsillar hypertrophy; and who have had adenotonsillectomy in the past.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Adenoid Size | 1 month
  Children's adenoid size will be estimated from lateral neck X-ray film based on the adenoidal/nasopharyngeal ratio and from nasal endoscopy based on the ratio of adenoid blocking posterior nostril. Lateral neck X-ray film and nasal endoscopy will be performed before and after the 1-month course.
Clinical responses including 9 symptoms (hard to awaken, witnessed apnea, breathing difficulties, snoring, sweating, mouth breathing, awakenings, restless sleep, wetting the bed) | 1 month
  Children's parents will be required to complete a questionnaire about 9 symptoms at diagnosis and after 1 month of therapy. Answers were scored are on a scale of 0 = never to 4 = most of the time.

SECONDARY OUTCOMES:
Tonsillar Size | 1 month
  estimation of oropharyngeal examination before and after the therapy.
Pediatric Sleep Questionnaire(PSQ) Score | 1 month
  Children's parents will be required to complete the PSQ questionnaire at diagnosis and after 1 month of therapy.
Obstructive Sleep Apnea Questionnaire(OSA-18) Score | 1 month
  Children's parents will be required to complete the OSA-18 questionnaire at diagnosis and after 1 month of therapy.
Polysomnography | 1 month
  Children's sleep will be estimated from polysomnography based on the apnea-hypopnea index, obstructive apnea index, time with oxygen saturation below 90% and minimum oxygen saturation value.
Lung function | 1 month
  Children's airway ventilation function will be estimated from lung function examination based on the FEV1/FVC value.
Nasal nitric oxide | 1 month
  Children's nasopharyngeal inflammation will be estimated based on the nasal nitric oxide value.

CONTACTS AND LOCATIONS:
Overall Officials: Shisheng Li, Ph.D., Principal Investigator — Department of Otolaryngology, Second Xiangya Hospital, Central South University
Locations (1):
- Department of Otolaryngology, Second Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thorsson L, Borga O, Edsbacker S. Systemic availability of budesonide after nasal administration of three different formulations: pressurized aerosol, aqueous pump spray, and powder. Br J Clin Pharmacol. 1999 Jun;47(6):619-24. doi: 10.1046/j.1365-2125.1999.00956.x. PMID 10383539
- [Background] Suman JD, Laube BL, Dalby R. Comparison of nasal deposition and clearance of aerosol generated by nebulizer and an aqueous spray pump. Pharm Res. 1999 Oct;16(10):1648-52. doi: 10.1023/a:1011933410898. No abstract available. PMID 10554112
- [Background] Goldbart AD, Greenberg-Dotan S, Tal A. Montelukast for children with obstructive sleep apnea: a double-blind, placebo-controlled study. Pediatrics. 2012 Sep;130(3):e575-80. doi: 10.1542/peds.2012-0310. Epub 2012 Aug 6. PMID 22869829
- [Background] Zhang Y, Lou H, Wang Y, Li Y, Zhang L, Wang C. Comparison of Corticosteroids by 3 Approaches to the Treatment of Chronic Rhinosinusitis With Nasal Polyps. Allergy Asthma Immunol Res. 2019 Jul;11(4):482-497. doi: 10.4168/aair.2019.11.4.482. PMID 31172717